CLINICAL TRIAL: NCT03722277
Title: Variable Resistance Training Versus Conventional Rubber Band Training: Effects on Functional Capacity and Strength in Patients With Osteoarthrosis of the Knee
Brief Title: Variable Resistance Training in Patients With Osteoarthrosis of the Knee
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College South Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Variable Load
Record Dates: First submitted 2018-10-18; First posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Variable load training (Experimental): The participants will be training two times per week in 10 weeks. Training will consist of variable load training in knee flexion- and extension.
  Training will be based on symptoms in isometric strength at five different angles of flexion- and extension.
  Interventions: Other: Variable load training
- Conventional strength training (Active Comparator): The participants will be training two times per week in 10 weeks. Training will consist of a training programme consisting of strength training with rubber bands for hip and knee.
  Interventions: Other: Conventional strength training

INTERVENTIONS:
Other: Variable load training — Based on symptoms/strength measured in an isometric maximum strength test at five different angles of knee flexion- and extension, participants will be training with variable load during both concentric and excentric phase of the dynamic movement. Initially participants will start at 40% of symptom limited isometric strength, this will increase to 50% during the training period.
  Arms: Variable load training
Other: Conventional strength training — Conventional strength training with rubber bands in knee flexion- and extension, additionally hip abduction- and adduction.
  Arms: Conventional strength training

SUMMARY:
This is a randomized controlled trial investigating the effect of variable load training in patients with knee osteoarthrosis.

The intervention will consist of resistance training with variable load in knee extension- and flexion. The control group will receive conventional strength training with rubber band.

Outcome measures will be the Knee Osteoarthrosis Outcome Score, functional capacity measured in a sit to stand test, 30m. pace walk and a 9 step stair climb test. Additionally isometric strength in knee flexion- and extension will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Knee pain and minimum three of the following
* >50 years
* morning stiffness < 30 min
* crepitation
* bone tenderness
* bone osteophytes
* absence of inflammation

Exclusion Criteria:

* Other causes of symptoms to the knee

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-10-22 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in self reported knee function | At baseline and 10 weeks follow up
  Knee Osteoarthrosis Outcome Score (100-0, 100 indicating no symptoms and 0 indicating extreme symptoms)

SECONDARY OUTCOMES:
Change in functional capacity | At baseline and 10 weeks follow up
  Sit to stand test
Change in isometric strength | At baseline and 10 weeks follow up
  Isometric strength in knee flexion- and extension
Change in functional capacity | At baseline and 10 weeks follow up
  30m pace walk
Change in functional capacity | At baseline and 10 weeks follow up
  9 step stair climb test

IPD SHARING:
Plan to Share IPD: No